CLINICAL TRIAL: NCT00197119
Title: Evaluate Persistence of Immune Response of GSK Biologicals' TWINRIX™ Vaccine Administered According to 0,6 Month Schedule Versus TWINRIX™ JUNIOR Administered According to 0,1,6 Month Schedule, in Subjects Aged 12-15 Years at Time of First Vaccine Dose
Brief Title: Long-Term Follow-Up Studies at Year 6, 7, 8, 9, 10: 2 Formulations of Combined Hepatitis A/B Vaccine Compared in Subjects Aged 12-15 Years
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 100566; 100567 (Other: GSK); 100568 (Other: GSK); 100569 (Other: GSK); 100570 (Other: GSK)
Record Dates: First submitted 2005-09-14; First posted 2005-09-20 (Estimated); Results first posted 2009-08-14 (Estimated); Last update posted 2017-04-20 (Actual); Status verified 2017-03

CONDITIONS: Hepatitis B; Hepatitis A
Keywords: Hepatitis B; TWINRIX™ Adult; Hepatitis A; TWINRIX™ Junior
MeSH Terms: conditions — Hepatitis B; Hepatitis A

ARMS (2):
- Group Twinrix Adult (Active Comparator): Subjects received Twinrix™ Adult (720/20) in a 0, 6 month schedule in the primary study.
  Interventions: Biological: Twinrix™ Adult
- Group Twinrix Junior (Active Comparator): Subjects received Twinrix™ Junior (360/10) in a 0, 1, 6 month schedule in the primary study.
  Interventions: Biological: Twinrix™ Junior

INTERVENTIONS:
Biological: Twinrix™ Adult — Intramuscular administration in the deltoid region (2 doses).
  Arms: Group Twinrix Adult
Biological: Twinrix™ Junior — Intramuscular administration in the deltoid region (3 doses).
  Arms: Group Twinrix Junior

SUMMARY:
To evaluate the persistence of anti-hepatitis A virus (anti-HAV) and anti-hepatitis B surface antigen (anti-HBs) antibodies up to 6, 7, 8, 9 and 10 years after administration of the first dose of the study vaccine.

DETAILED DESCRIPTION:
Open, randomized, long-term antibody persistence studies. Immune persistence was compared between subjects who received one of the two formulations of GlaxoSmithKline Biologicals' combined hepatitis A and hepatitis B vaccine according to a two-dose or three-dose schedule. These long-term follow-up studies involved taking blood samples at approximately 6, 7, 8, 9 and 10 years after the primary vaccination of combined hepatitis A and B vaccine, to assess antibody persistence and a retrospective safety follow-up.

The Protocol Posting has been updated in order to comply with the FDA Amendment Act, Sep 2007.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and female volunteers vaccinated in study HAB-084.
* Written informed consent obtained from the subject before the blood sampling visit of each year.

Exclusion Criteria:

• none

Ages: 12 Years to 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 244 (Actual)
Dates: Start 2004-05; Primary Completion 2004-06 (Actual); Study Completion 2004-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (2):
- GSK Investigational Site, Brussels, Belgium
- GSK Investigational Site, Hradec Králové, Czechia

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Background] Beran J, Kervyn D, Wertzova V, Hobzova L, Tichy P, Kuriyakose S, Leyssen M, Jacquet JM. Comparison of long-term (10 years) immunogenicity of two- and three-dose regimens of a combined hepatitis A and B vaccine in adolescents. Vaccine. 2010 Aug 23;28(37):5993-7. doi: 10.1016/j.vaccine.2010.06.104. Epub 2010 Jul 15. PMID 20637766
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Individual Participant Data Set: 100566 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register. The results of this study 100566 are summarised with studies 100567, 100568, 100569, and 100570 on the GSK Clinical Study Register.
- Available data/document: Clinical Study Report: 100566 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 100566 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 100566 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 100566 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 100566 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Recruitment Details: At the time of initiation of the long-term follow-up study, the investigators contacted the subjects who had consented to participate in the long-term follow-up studies. At each subsequent visit, subjects who were present at the previous long-term blood sampling time points were contacted again.
Period: Year 6
Arm/Group | Group Twinrix Junior | Group Twinrix Adult
Started | 126 | 118
Completed | 126 | 118
Not Completed | 0 | 0
Period: Year 7
Arm/Group | Group Twinrix Junior | Group Twinrix Adult
Started | 122 (4 subjects who participated in the Year 6 follow-up time point did not return for this time point.) | 114 (4 subjects who participated in the Year 6 follow-up time point did not return for this time point.)
Completed | 122 | 114
Not Completed | 0 | 0
Period: Year 8
Arm/Group | Group Twinrix Junior | Group Twinrix Adult
Started | 122 | 115 (One additional subject (compared to Year 7) participated in the current follow-up time point.)
Completed | 122 | 115
Not Completed | 0 | 0
Period: Year 9
Arm/Group | Group Twinrix Junior | Group Twinrix Adult
Started | 121 (One subject participating in the Year 8 time point did not return for the current time point.) | 114 (One subject participating in the Year 8 time point did not return for the current time point.)
Completed | 121 | 114
Not Completed | 0 | 0
Period: Year 10
Arm/Group | Group Twinrix Junior | Group Twinrix Adult
Started | 120 (One subject participating in the Year 9 time point did not return for the current time point.) | 108 (Six subjects participating in the Year 9 time point did not return for the current time point.)
Completed | 120 | 108
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group Twinrix Junior | Group Twinrix Adult | Total
Number analyzed (Participants) | 126 | 118 | 244
Age, Continuous [Mean (Standard Deviation); unit: years] — Subjects' mean age at Year 6, the time of first enrollment into the long-term follow-up phase of the study.
  years | 19.4 (1.04) | 19.4 (1.12) | 19.4 (1.08)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 62 | 61 | 123
  Male | 64 | 57 | 121

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With Anti-hepatitis A Virus (HAV) Antibody Concentrations Above the Cut-off Value
Description: Anti-HAV antibody concentration cut-off value assessed was ≥ 15 milli-International Units per milliliter (mIU/mL).
Time Frame: Year 6, 7, 8, 9 and 10 after the first vaccine dose of a two-dose or three-dose primary vaccination
Population: Analysis was performed on the Long Term According To Protocol (ATP) cohort for immunogenicity, which included all subjects for whom serology results were available for a particular blood sampling visit.
Measure: Number; unit: subjects
Arm/Group | Group Twinrix Junior | Group Twinrix Adult
Number analyzed (Participants) | 113 | 100
subjects
  Year 6 (n=113, 100) | 113 | 100
  Year 7 (n= 105, 92) | 105 | 92
  Year 8 (n= 104, 93) | 104 | 93
  Year 9 (n= 103, 90) | 103 | 90
  Year 10 (n= 100, 77) | 100 | 77

2. Primary Outcome: Number of Subjects With Anti-Hepatitis B Surface Antigen (HBs) Antibody Concentrations Above the Cut-Off Value
Description: Anti-HBs antibody concentration cut-off value assessed was ≥ 3.3 mIU/mL.
Time Frame: Year 6, 7, 8, 9 and 10 after the first vaccine dose of a two-dose or three-dose primary vaccination
Population: Analysis was performed on the ATP cohort for immunogenicity, which included all subjects for whom serology results were available for a particular blood sampling visit.
Measure: Number; unit: subjects
Arm/Group | Group Twinrix Junior | Group Twinrix Adult
Number analyzed (Participants) | 113 | 100
subjects
  Year 6 (n= 113, 100) | 100 | 93
  Year 7 (n= 105, 92) | 98 | 85
  Year 8 (n= 104, 93) | 96 | 84
  Year 9 (n= 103, 90) | 96 | 86
  Year 10 (n= 101, 78) | 97 | 75

3. Primary Outcome: Serious Adverse Events (SAE) Causally Related to Primary Vaccination or Related to Hepatitis A or B Infection or Related to Study Participation (Blood Sampling)
Description: An SAE is any untoward medical occurrence that:
  results in death, is life-threatening, requires hospitalization or prolongation of existing hospitalization, results in disability/ incapacity, is a congenital anomaly/birth defect in the offspring of a study subject, or may evolve into one of the outcomes listed above.
Time Frame: From Year 6 through to Year 10
Measure: Number; unit: subjects
Arm/Group | Group Twinrix Junior | Group Twinrix Adult
Number analyzed (Participants) | 126 | 118
subjects | 0 | 0

ADVERSE EVENTS:
Time Frame: From Year 6 through to Year 10.
Description: Other (non-serious) adverse event data was not collected during this long-term follow-up phase of the study.
Arm/Group | Group Twinrix Junior | Group Twinrix Adult
Serious Adverse Events (participants affected / at risk) | 0/126 | 0/118
Other Adverse Events (participants affected / at risk) | 0/126 | 0/118

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.